CLINICAL TRIAL: NCT01604369
Title: Cryoablation as Standard Treatment of Atrial Flutter - Long Term Efficacy and Patient Content
Brief Title: Cryoablation as Standard Treatment of Atrial Flutter
Acronym: CASTAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Jensen-Urstad, Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KS1
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Atrial Flutter
Keywords: Atrial flutter; Cryoablation; Cavotricuspid isthmus; Visual analogue scale
MeSH Terms: conditions — Atrial Flutter | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryoablation (Experimental)
  Interventions: Procedure: Medtronic Freezor Max Cardiac Cryoablation Catheter

INTERVENTIONS:
Procedure: Medtronic Freezor Max Cardiac Cryoablation Catheter — Cryoablation is performed using a sequential application technique point-by-point from the tricuspid annulus to the inferior vena cava. Ablation is performed at a target temperature of -80 ºC. Each application will last for 240 seconds.
  Other Names: Cryoablation; CTI ablation

SUMMARY:
The hypothesis of the present study is to evaluate cryoablation(cooling of the tissue) as standard therapy of common atrial flutter,focusing on efficacy, feasibility, procedure time, and patient content.

The purpose of this study is to determine whether cryoablation, performed only by operators experienced in cryothermic ablation is effective and safe in the treatment of atrial flutter.

DETAILED DESCRIPTION:
Atrial flutter (AFL), a common atrial tachyarrhythmia may cause significant symptoms and serious adverse effects including embolic stroke, myocardial ischemia and congestive heart failure. Currently, radiofrequency (RF) catheter ablation of the cavotricuspid isthmus (CTI) is considered first-line therapy for treatment of CTI-dependent AFL. However, RF ablation of the CTI is associated with significant pain during lesion delivery. Furthermore, RF ablation can potentially injure cardiac structures adjacent to the CTI such as the AV node, tricuspid valve and right coronary artery. RF ablation can also lead to steam pops, cardiac tamponade and fatal complications have also been reported in association with CTI-ablation. Ablation using cryothermal energy (Cryo) has several potential advantages over RF ablation including greater catheter stability due to adherence to myocardial tissue during applications, reduced risk of thrombus formation, systemic embolization, and lower risk of myocardial perforation due to preservation of tissue architecture.

The investigators have in a prospective randomized, single centre study (CRAFT) investigated efficacy and safety of RF versus Cryo for atrial flutter, and showed that cryoablation is as effective as RF ablation in the short and long term. The patients perceived significantly less pain and required significantly lower doses of analgesia and sedation during cryoablation compared to RF ablation. The study was powered for non-inferiority with 75 patients in each group.

The objective of the present study is to expand the findings from the CRAFT study in a larger cohort of patients, letting only operators experienced in cryothermic CTI ablation use Cryo as standard therapy focusing on efficacy, feasibility, procedure time, and patient content.

To perform an ablation within the study, the electrophysiologist must have a previous experience of a minimum of 25 cryoablations of atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients referred to our institution for ablation therapy of ECG-documented, typical CTI dependent AFL.
* Patients above the age of 18 having symptomatic CTI-dependent AFL documented on a 12-lead ECG with typical ECG appearance of negative saw tooth waves in the inferior limb leads and positive deflections in V1 or positive saw tooth waves in the inferior limb leads and negative deflections in V1.
* Patients with a history of atrial fibrillation will only be included if they have predominant atrial flutter under chronic treatment with class I or III antiarrhythmic agents.

Exclusion Criteria:

1. prior ablation for AFL;
2. atrial flutter related to recently undergone surgery, hyperthyroidism or other severe disease;
3. inability to adhere with the study protocol;
4. pregnancy;
5. predominant atrial fibrillation; and
6. for patients with persistent atrial flutter contraindication to warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | One year after intervention
  Clinical success defined as the freedom from atrial flutter evaluated at the 12-month follow-up.

SECONDARY OUTCOMES:
Safety | During and up to one year after intervention
  The secondary endpoints will be acute ablation success defined as bidirectional CTI-block, safety assessed by the rate of periprocedural complications, procedure and fluoroscopy times and the level of pain experienced by the patient during the ablation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jensen-Urstad, Professor, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden